CLINICAL TRIAL: NCT06287268
Title: Revolade Tablets Specified Drug-use Survey (Pediatric Aplastic Anemia Naive to Treatment With Anti-thymocyte Immunoglobulin, CETB115G1401)
Brief Title: Revolade Tablets Specified Drug-use Survey
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CETB115G1401
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Aplastic Anemia
Keywords: NIS; Pediatric Aplastic Anemia; AA; Revolade Tablets; eltrombopag; Drug-use Survey
MeSH Terms: conditions — Anemia, Aplastic | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- eltrombopag: ATG treatment naïve pediatric patients with AA in routine clinical practice
  Interventions: Other: eltrombopag

INTERVENTIONS:
Other: eltrombopag — This is an observational study. There is no treatment allocation. After confirming that patients are fulfilling the eligibility criteria, patients will be registered in this survey.

SUMMARY:
This is a multicenter, single-arm, non-interventional study (NIS) to confirm the safety and efficacy of eltrombopag in Anti-Thymocyte Globulin (ATG) treatment naive pediatric patients with aplastic anemia (AA).

DETAILED DESCRIPTION:
The objective of this survey is to confirm the safety and efficacy of eltrombopag in ATG treatment naive pediatric patients with AA. Eltrombopag should be administered according to the dosage and administration specified in the latest version of the package insert. The observation period is 1 year (364 days) from the start of treatment with this product, regardless of whether treatment with eltrombopag is continued or not. However, if hematopoietic stem cell transplantation is performed within 1 year after the start of treatment with eltrombopag, the observation period shall be until the date of hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose legally acceptable representative has given written consent for cooperation in this survey prior to enrollment in this survey
* Patients aged ≥ 6 years and < 18 years at the start of treatment with eltrombopag
* Pediatric patients with AA who receive eltrombopag for the first time in combination with ATG after the approval of additional dosage and administration for "ATG-naïve pediatric patients with AA"

Exclusion Criteria:

* Patients who have received ATG without concomitant use of eltrombopag
* Patients with congenital AA
* Patients with suspected or confirmed diagnosis of myelodysplastic syndrome (MDS) at the start of treatment with eltrombopag
* Patients who have received any drug products containing the same ingredient as eltrombopag (including investigational products)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The survey will be conducted in pediatric patients with Aplastic anemia (AA) who receive eltrombopag for the first time in combination with ATG after the approval of additional dosage and administration for "ATG-naïve pediatric patients with AA."
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2029-03-28 (Estimated); Study Completion 2029-03-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence of serious adverse events | Up to 1 year
  Occurrence of serious adverse events to be provided

SECONDARY OUTCOMES:
Occurrence of adverse events and adverse drug reactions leading to treatment discontinuation | Up to 1 Year
  Occurrence of adverse events and adverse drug reactions leading to treatment discontinuation to be provided
Occurrence of adverse events and adverse drug reactions applicable to safety specifications (hepatic dysfunction and hematopoietic malignancies) | Up to 1 year
  Occurrence of adverse events and adverse drug reactions applicable to safety specifications (hepatic dysfunction and hematopoietic malignancies)
Occurrence of clonal evolution | Up to 1 year
  Occurrence of clonal evolution [cytogenetic abnormalities, myelodysplastic syndrome (MDS), Acute Myeloid Leukemia (AML), and paroxysmal nocturnal hemoglobinuria (PNH)]
Hematologic response status | Up to 1 year
  Hematologic response status to be provided
Change over time from baseline in platelet count | Baseline, 1 year
  Change over time from baseline in platelet count to be provided
Change over time from baseline in hemoglobin | Baseline, 1 year
  Change over time from baseline in hemoglobin to be provided
Change over time from baseline in neutrophil count | Baseline, 1 year
  Change over time from baseline in neutrophil count to be provided
Change over time from baseline in reticulocyte count | Baseline, 1 year
  Change over time from baseline in reticulocyte count to be provided
Change over time from baseline in transfusion dependence | Baseline, 1 year
  Change over time from baseline in transfusion dependence to be provided
Change over time from baseline in transfusion volume | Baseline, 1 year
  Change over time from baseline in transfusion volume to be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Shimajiri-Gun, Okinawa
  - Novartis Investigative Site, Izumi, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama

IPD SHARING:
Plan to Share IPD: No